CLINICAL TRIAL: NCT07044882
Title: Evaluation of the Hydrodynamic Piezoelectric Technique in Internal Sinus Lift With Simultaneous Implant Placement (A Randomized Controlled Clinical Trial)
Brief Title: Hydrodynamic Piezoelectric Technique in Internal Sinus Lift
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-H-0165-D-M-0752
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Maxillary Sinus Lift; Osteotome
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional osteotome technique (Active Comparator)
  Interventions: Procedure: conventional osteotome technique
- osteotome with hydrodynamic piezoelectric (Experimental)
  Interventions: Procedure: Hydrodynamic Piezoelectric technique

INTERVENTIONS:
Procedure: conventional osteotome technique — Patients indicated for internal sinus lifting with simultaneous implant placement, where sinus elevation is conducted with regular manual osteotomes.
  Other Names: Control group
  Arms: conventional osteotome technique
Procedure: Hydrodynamic Piezoelectric technique — Patients indicated for internal sinus lifting with simultaneous implant placement, where sinus elevation is conducted with Hydrodynamic Piezoelectric technique.
  Arms: osteotome with hydrodynamic piezoelectric

SUMMARY:
Background: The use of hydrodynamic piezoelectric techniques for trans crestal / internal sinus lift with simultaneous implant placement has gained popularity as a safe and minimally invasive technique for managing the posterior edentulous maxilla, particularly in cases with sinus pneumatization. This method offers a controlled elevation of the Schneiderian membrane while reducing the risk of perforation compared to conventional techniques. Additionally, it minimizes postoperative discomfort and oedema, leading to better acceptance and satisfaction by the patients. In contrast to traditional osteotome tapping procedures, the hydrodynamic piezoelectric technique enhances surgical outcomes while preserving vital anatomical structures, making it a superior alternative in implant dentistry. This study aims to evaluate the use of the hydrodynamic piezoelectric technique in internal sinus lifting with simultaneous implant placement in comparison to the conventional osteotome technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients with edentulous free end or bounded posterior maxilla that require implant supported restoration.
* Patients indicated to internal sinus lifting, where insufficient residual alveolar bone height from the alveolar crest to the floor of the maxillary sinus is found.
* Patients with residual alveolar bone height that ranges from 5-7 mm according to the tomographic radiographic examination.
* A good standard of oral hygiene.

Exclusion criteria:

* Patients with residual alveolar bone height less than 5 mm according to the tomographic radiographic examination.
* Patients with residual alveolar bone height more than 8 mm according to the tomographic radiographic examination, which is not indicated to sinus lifting.
* Patient with active sinus infection or sinus pathology.
* History of Oral or intravenous bisphosphonate therapy or any treatments with other medications that may interfere with bone metabolism within the past 12 months.
* Heavy smokers.
* Medically compromised patients that are burdened with systemic conditions that contradicts implant placement and interfere with wound healing.

Exclusion Criteria:

-

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain scores | at 7, 14, and 21 days
  Pain will be evaluated, using visual analogue scale (VAS) as follows:
  (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe).
Change in wound healing | at 7, 14, and 21 days
  The wound healing will be assessed based on the Modified Healing Index. The Wound Healing Index (WHI) evaluates preimplant soft tissue wound healing with scores from 1 to 3. On this scale, a score of 1 indicates ordinary healing with the absence of gingival edema, erythema, suppuration, patient discomfort, and flap dehiscence. A score of 2 indicates ordinary healing with slight gingival edema, erythema, patient discomfort, and flap dehiscence, but no suppuration and a score of 3 corresponds to poor wound healing with significant gingival edema, erythema, patient discomfort, suppuration, and flap dehiscence, or any suppuration
change in implant stability | baseline and 6 months
  Implant Stability Quotient (ISQ) will be measured during the operative stage, while the secondary stability quotient will be measured 6-months post-operative during the prosthetic phase preparation using Ostell device.

SECONDARY OUTCOMES:
Change in Alveolar Process height gain | baseline and 6 months
  The baseline residual alveolar bone height will be measured in the preoperative scan from the alveolar crest to the maxillary sinus floor. Immediate postoperative alveolar bone height will be measured to outline the effectiveness of sinus membrane elevation using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry clinics, Beirut Arab University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No